CLINICAL TRIAL: NCT05500482
Title: Vellore Typhoid Vaccine Impact Trial
Acronym: VEVACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University College, London (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Jacob John, Professor, Christian Medical College, Vellore, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14247[INTERVEN]
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Typhoid Fever
Keywords: typhoid conjugate vaccine; cluster randomised trial; Enteric Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The control arm will not receive a vaccine, however the investigator and the outcome assessors will be trained not to seek history of vaccination. The clusters selected for vaccination and their boundaries will not be accessible to the investigators and outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccinated arm (Experimental): Typhoid Conjugate Vaccine (TyphiBEV) 0.5 ml as a single dose given intramuscularly to consenting, eligible residents of vaccine clusters
  Interventions: Biological: Typhoid conjugate Vaccine
- Control arm (No Intervention): No vaccination in the control clusters

INTERVENTIONS:
Biological: Typhoid conjugate Vaccine — TyphiBEV is a clear colourless monovalent vaccine containing 25 µg of Typhoid Vi polysaccharide manufactured using the Citrobacter freundii sensu lato3056 (Vi) and is conjugated to CRM 197 as a carrier protein. Sodium chloride and Phosphate buffer are used as a buffering agent in the vaccine formulation with 2-Phenoxyethanol as a preservative.
  Other Names: TyphiBEV
  Arms: Vaccinated arm

SUMMARY:
This cluster randomised trial will examine the impact of introducing TyphiBEV, a typhoid conjugate vaccine licensed in India, on the incidence of typhoid fever in a high burden urban setting in South India.

DETAILED DESCRIPTION:
TyphiBEV®, a typhoid conjugate vaccine from Biological E, has been licensed by the Central Drugs Standard Control Organaisation in India based on immunogenicity and safety data. A similar typhoid conjugate vaccine has been demonstrated in large clinical trials to provide 80% vaccine efficacy in Nepal and Bangladesh. The TyphiBEV® has not been similarly evaluated. The demonstration of the impact of a city-scale typhoid conjugate vaccine introduction on the burden of typhoid will aid policy decisions on the use of typhoid conjugate vaccines in the national immunisation program.

After written informed consent, the investigators will establish stimulated passive surveillance in 72,000 individuals between 1 and 30 years of age within the Vellore Demographic Surveillance System to determine the incidence of blood-culture confirmed typhoid fever. Thirty-six thousand surveillance participants between 1 year and 30 years residing in the 30 clusters (areas) randomised to receive the vaccine will receive the vaccine at the beginning of the trial. Those in other areas will receive the same at the end of two years. Using a stimulated passive surveillance approach, those with acute febrile illness will be encouraged to visit study surveillance hospitals. Participants will be evaluated for blood-culture confirmed typhoid fever if they are eligible. The incidence of typhoid among those living in areas assigned to vaccination compared to those whose residence is in areas not designated for vaccination will be used to calculate the impact of the vaccine on disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Consent

  * For adults, 18 years and over - they must be willing and competent to provide informed consent
  * For those aged under 18 years, the parent/guardian is willing and competent to provide informed consent, and if the participant is 11 to 18 years of age, informed assent will also be sought,
* Age:

  * Between 1 and 30 years (i.e., up to 29 years 364 days) at time of recruitment into the surveillance
  * Currently living within the study catchment area with no plans to leave the study area in the next 24 months

Exclusion Criteria:

* For fever surveillance

  o Medical reasons that prevent the participant from complying with study requirements including follow up and testing during illness
* For vaccination

  * Has received a typhoid vaccine in the previous three years
  * Is known to have an allergy to any vaccine component
  * Nursing mothers, Pregnancy or planning pregnancy around vaccination
  * Receipt of any other vaccine in the past 30 days (temporary exclusion)
  * Febrile illness in the 24 hours before vaccination (temporary exclusion)

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total effect | at 24 months of follow up beginning 28 days after vaccine introduction in vaccine clusters.
  Number of blood culture confirmed typhoid fever episodes in vaccinated participants from vaccine clusters compared to the number of blood culture confirmed typhoid fever episodes in unvaccinated participants from non-vaccine clusters

SECONDARY OUTCOMES:
Overall effect | at 24 months of follow up beginning 28 days after vaccine introduction in vaccine clusters.
  The number of blood culture confirmed typhoid fever episodes in participants from vaccine clusters compared to the number of blood culture confirmed typhoid fever episodes in participants from non-vaccine clusters
Effect in children 1 to 14 years | at 24 months of follow up beginning 28 days after vaccine introduction in vaccine clusters.
  The number of blood culture confirmed typhoid fever episodes in vaccinated children between 1 year and 14 years and 364 days from vaccine clusters compared to the number of blood culture confirmed typhoid fever episodes in unvaccinated children between 1 year and 14 years and 364 days from non-vaccine clusters
Effect on all febrile illness requiring healthcare visits | at 24 months of follow up beginning 28 days after vaccine introduction in vaccine clusters.
  The number of febrile illness episodes where healthcare is sought among vaccinated participants from vaccine clusters compared to unvaccinated participants from non-vaccine clusters
Safety outcomes | Seven days after vaccine receipt
  The number and description of solicited and non-solicited adverse events reported within the first seven days after vaccination in the safety subset of vaccine recipients

OTHER OUTCOMES:
Indirect effect | at 24 months of follow up beginning 28 days after vaccine introduction in vaccine clusters.
  The number of blood culture confirmed typhoid fever episodes in unvaccinated participants from vaccine clusters compared to the number of blood culture confirmed typhoid fever episodes in unvaccinated participants from non-vaccine clusters
Effect on hospitalised typhoid fever | at 24 months of follow up beginning 28 days after vaccine introduction in vaccine clusters.
  The number of blood culture confirmed typhoid fever episodes in hospitalised participants who have been vaccinated compared to the number of blood culture confirmed typhoid fever episodes in hospitalised participants who have not been vaccinated

CONTACTS AND LOCATIONS:
Overall Officials: Jacob John, MD PhD, Principal Investigator — Christian Medical College, Vellore, India; Gagandeep Kang, MD PhD, Study Chair — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College Vellore, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual level data as permitted by the local law will be made available on Mendeley Data. Access to data will be possible by writing to the vevact@tympact.in on or after 31 Dec 2025
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of data lock at the end of the trial and for a period of five years thereafter
Access Criteria: Upon providing a draft hypothesis and analysis plan